CLINICAL TRIAL: NCT00592033
Title: Effect of Ambulatory Oxygen in Normoxaemic COPD Patients Who Desaturate During Exercise. A Randomised Placebo Controlled Trial of Patients Who Participate in Pulmonary Rehabilitation
Brief Title: Effect of Oxygen in Normoxaemic COPD Patients Who Desaturate During Exercise
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Danish Lung Association (Other)
Responsible Party: Principal Investigator, Thomas Ringbaek, Senior Consultant, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-41-0569
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: COPD
Keywords: COPD oxygen; COPD rehabilitation; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): Rehabilitation, no supplemental oxygen
- 1 (Experimental): Rehabilitation plus supplemental oxygen
  Interventions: Other: oxygen from a portable concentrator

INTERVENTIONS:
Other: oxygen from a portable concentrator — 2 l/minute during exercise
  Arms: 1

SUMMARY:
In COPD patients with desaturation during exercise, several studies have shown an acute beneficial effect of supplemental oxygen. Therefore, both the British Thoracic Society and the American Thoracic Society guidelines recommend supplemental oxygen to patients who desaturate >4% and to below 88-90%. However, long-term studies have not been able to support this intervention. In this study of COPD patients, who desaturate and participate in a 7-week pulmonary rehabilitation programme, we examine the effect of supplemental oxygen on exercise tolerance, health status, and exacerbation rates. In a randomised design patients trained either with room air or with 2 litres oxygen per minute from a portable oxygen concentrator. All patients were asked to exercise every day for 30 minutes.

DETAILED DESCRIPTION:
In COPD patients with desaturation during exercise, several studies have shown an acute beneficial effect of supplemental oxygen. Therefore, both the British Thoracic Society and the American Thoracic Society guidelines recommend supplemental oxygen to patients who desaturate >4% and to below 88-90%. However, long-term studies have not been able to support this intervention. In this study of COPD patients, who desaturate and participate in a 7-week pulmonary rehabilitation programme, we examine the effect of supplemental oxygen. Using a randomised design, patients trained either with room air (control) or with 2 litres oxygen per minute from a portable oxygen concentrator. All patients were asked to exercise every day for 30 minutes.

Primary effect parameters:

endurance shuttle walk time at baseline, 7 weeks (after intensive supervised rehabilitation), 3 months (after maintenance training twice a month), and after 6 months.

Secondary effect parameters:

St. George Respiratory Questionnaire (health status); usage of oxygen, exacerbations requiring medical treatment, hospitalisation and mortality in the same periods.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* participate in a 7-weeks pulmonary rehabilitation programme
* desaturate >4% to less than 90% during endurance shuttle walk test

Exclusion Criteria:

* long-term oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Shuttle walk (endurance time) | 7 week, 3 and 6 months

SECONDARY OUTCOMES:
St. George Respiratory Questionnaire | 7 week, 3 and 6 months
Usage of oxygen concentrator (Spent time according to the meter) | 7 weeks, 3 and 6 months
Exacerbations requiring medical treatment (prednisolone or antibiotics) | 7 weeks, 3 and 6 months
Hospitalisation | 7 weeks, 3 and 6 months
Mortality | 7 weeks, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Ringbaek, doctor, Principal Investigator — Hvidovre Hospital, University hospital, Cardio-pulmonary depart.
Locations (1):
- University Hospital, Hvidovre, Cardio-pulmonary depart., Hvidovre, Denmark